CLINICAL TRIAL: NCT02818725
Title: Intensified Methotrexate, Vinblastine, Doxorubicin and Cisplatin +/-Panitumumab as First-line Treatment of Advanced Urothelial Carcinoma in Patients Without Harvey Nor Kirsten Rat Sarcoma Viral Oncogene Homolog Mutations. Phase II Study
Brief Title: I-MVAC +/- Panitumumab as First-line Treatment of Advanced Urothelial Carcinoma Without H-Ras Nor K-Ras Mutations
Acronym: GETUG-AFU19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-AFU 19/0903; 2009-011882-10 (EudraCT Number)
Record Dates: First submitted 2011-11-29; First posted 2016-06-30 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Infiltrating Urothelial Carcinoma; KRAS Gene Mutation
MeSH Terms: interventions — Drug Therapy; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): Intensified- Methotrexate Vinblastin Doxorubicin Cisplatin
  Interventions: Drug: Chemotherapy
- Arm B: chemotherapy + panitumumab (Experimental): Intensified- Methotrexate Vinblastin Doxorubicin Cisplatin +/- panitumumab
  Interventions: Drug: Chemotherapy; Drug: Panitumumab

INTERVENTIONS:
Drug: Chemotherapy — METHOTREXATE: 30 mg/m² on day 1 VINBLASTINE: 3 mg/m² on day 2 DOXORUBICIN: 30 mg/m² on day 2 CISPLATIN: 70 mg/m² on day 2
  Other Names: Intensified-Methotrexate Vinblastine Doxorubicin Cisplatin; I-MVAC
Drug: Panitumumab — PANITUMUMAB: 6 mg/kg on day 2
  Arms: Arm B: chemotherapy + panitumumab

SUMMARY:
OBJECTIVES OF THE TRIAL

Primary objective

Evaluation of efficacy in terms of progression-free survival at 9 months of the combination of intensified methotrexate, vinblastine, doxorubicin and cisplatin with or without panitumumab as first-line treatment of advanced urothelial carcinoma in patients without Harvey nor Kirsten rat sarcoma viral oncogene homolog mutations.

Secondary objectives

* To assess toxicity
* To assess response rate
* To assess overall survival
* To assess time to progression
* To study the correlation between response rate, time to progression, overall survival and biological parameters

ELIGIBILITY:
Inclusion Criteria:

1. Primary tumour of the bladder or upper urinary tract
2. Histologically confirmed infiltrating urothelial carcinoma (epidermoid and/or glandular forms are accepted)
3. Patients without Harvey and Kirsten-rat sarcoma viral oncogene homolog mutations
4. Advanced disease defined by a locally advanced stage (T4 and/or N+) ineligible for surgical resection, or a metastatic stage (M1)
5. Patients with at least 1 evaluable lesion as per Response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)
6. 18 ≤ age ≤ 75 years
7. General condition 0 or 1 as per the WHO scale
8. Absence of previous chemotherapy for advanced disease (chemotherapy with gemcitabine and platinum salt delivered as an adjuvant is accepted if this ended more than a year ago)
9. Haematological function: Haemoglobin >11 g/dl, neutrophils ≥1500/mm³, platelets ≥100,000/mm³
10. Liver function: Grade* 0 Aspartate aminotransferase and Alanine aminotransferase (< grade* 3 for liver metastases), grade* 0 alkaline phosphatases, normal bilirubin
11. Renal function: calculated (or measured) creatinine clearance >60 ml/min
12. Patients covered by a social security scheme
13. Patient having read the information sheet and signed the informed consent form.

Exclusion Criteria:

1. Pure adenocarcinoma or pure epidermoid carcinoma or mixed or pure small-cell neuroendocrine carcinoma
2. Previous treatment with one of the following molecules: methotrexate, vinblastine, doxorubicin or Epidermal Growth Factor inhibitor
3. History of interstitial pneumonitis or pulmonary fibrosis
4. History of cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, uncontrolled serious cardiac arrhythmia) in the year prior to randomisation (≤1 year)
5. Ventricular ejection fraction <50%
6. Blood calcium and/or magnesium ≥ grade* 1
7. History of cancer in the 5 years prior to entry in the trial other than basal cell skin cancer or in situ epithelioma of the cervix,
8. Treatment with radiotherapy for analgesic purposes (unless treatment was discontinued at least 15 days prior to inclusion in the trial)
9. Potential allergy to panitumumab
10. Male or female patients not agreeing to use an effective method of contraception throughout the duration of treatment and for 6 months after treatment discontinuation
11. Pregnant women, or female subjects liable to become pregnant or currently breast-feeding,
12. Patient already included in another therapeutic trial on an investigational medicinal product,
13. Persons deprived of their freedom or under judicial protection (including guardianship),
14. Unable to receive medical follow-up during the trial owing to geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Time to progression | 9 months
  Progression-Free Survival at 9 months post-treatment

SECONDARY OUTCOMES:
Toxicities assessment | 24 months
  toxicity (CTC AE v4.0) after end of treatment
Evaluation of response | 24 months
  Recist 1.1
Evaluation of overall survival | 24 months
Evaluation of time to progression | 24 months

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Hopital Henri Mondor, Créteil
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Alexis Vautrin, Nancy
  - Centre Rene Gauducheau, Nantes
  - Chu de Nimes, Nîmes
  - Institut Curie, Paris
  - Diaconesses - Croix St Simon, Paris
  - Pitie Salpetriere, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Cancerologie de La Loire, Saint-Priest-en-Jarez
  - Hopitaux Universitaires, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes